CLINICAL TRIAL: NCT04631471
Title: Regeneration in Cervical Degenerative Myelopathy - a Multi-centre, Double-blind, Randomised, Placebo Controlled Trial Assessing the Efficacy of Ibudilast as an Adjuvant Treatment to Decompressive Surgery for Degenerative Cervical Myelopathy
Brief Title: Regeneration in Cervical Degenerative Myelopathy
Acronym: RECEDE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Mark R Kotter, Chief Investigator, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCTU0178; 2017-004856-41 (EudraCT Number); 213009 (Registry Identifier: IRAS)
Record Dates: First submitted 2020-07-09; First posted 2020-11-17 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Myelopathy; Spinal Cord Diseases
Keywords: Degenerative; Cervical; Myelopathy
MeSH Terms: conditions — Spinal Cord Diseases | interventions — ibudilast

STUDY DESIGN:
Intervention Model Description: Placebo controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ibudilast (Active Comparator): Increasing dose of Ibudilast up to 100mg/day for up to 10 weeks prior to cervical decompressive surgery and up to 24 weeks after cervical decompressive surgery
  Interventions: Drug: Ibudilast; Procedure: Cervical decompressive surgery
- Placebo (Placebo Comparator): Increasing dose of matched placebo containing mannitol instead of ibudilast up to 10 pills/day for up to 10 weeks prior to cervical decompressive surgery and up to 24 weeks after cervical decompressive surgery
  Interventions: Procedure: Cervical decompressive surgery; Drug: Matching placebo

INTERVENTIONS:
Drug: Ibudilast — Increasing dose of ibudilast from 60mg/6 capsules per day to 100mg/10 capsules per day to be started up to 10 weeks prior to surgery. Treatment will continue up to 24 weeks after surgery. Maximum treatment period will be of 34 weeks.
  Arms: Ibudilast
Procedure: Cervical decompressive surgery — Surgical decompression of degenerate cervical myelopathy
Drug: Matching placebo — Increasing dose of matching placebo from 6 capsules per day to 10 capsules per day to be started up to 10 weeks prior to surgery. Treatment will continue up to 24 weeks after surgery. Maximum treatment period will be of 34 weeks.
  Arms: Placebo

SUMMARY:
Degenerative (wear and tear arthritis of the spine) Cervical (concerning the neck) Myelopathy (injury to the spinal cord), DCM, is the most common spinal cord disorder of adulthood. In DCM, arthritis of the spine causes compression of the spinal cord.

The symptoms of DCM are often mistaken for natural consequences of ageing, including numb and clumsy hands, loss of coordination, imbalance, bladder and bowel problems. The weakness can progress to severe paralysis. Every year approximately 4 individuals in 100,000 undergo surgery for DCM; however, many more individuals are thought to suffer from DCM.

The main treatment for DCM is surgery. The aim of surgery is to create space and remove the compression of the spinal cord. This is known to prevent further injury. Unfortunately, the post-operative improvements are often incomplete and many patients remain severely disabled. Improving outcome after surgery represents an important unmet clinical need.

Clinical and preclinical findings indicate that the drug Ibudilast can stimulate neuroprotective and regenerative processes in the spinal cord. Ibudilast is well-tolerated and used to treat asthma and post-stroke dizziness in Japan and is currently being investigated for use in treating other neurological diseases.

This study will investigate whether daily oral administration of Ibudilast for a maximum of 34 weeks can improve hand function, strength, balance, urinary problems and reduce pain.

The study will initially be conducted at three sites in the UK, with more sites added as necessary. Individuals between 18-80 years old, diagnosed with DCM and scheduled for an operation for the first time will be invited to participate in the trial. The study will entail patient questionnaires and clinical assessments before surgery, shortly after surgery and 3, 6, and 12 months after surgery. Moreover, patients will undergo MRI scans pre-operatively and at 6-months postoperatively to determine whether the treatment was successful.

DETAILED DESCRIPTION:
DCM is a common, disabling disease. It is also a major cause of gait disturbance and imbalance in the elderly. As a consequence, DCM contributes to reduced mobility and frailty. NHS England recognises 1) reducing premature mortality and 2) enhancing quality of life for people with long-term conditions as important. DCM patients are at risk of recurrent falls, which is a major concern. In fact, a study investigating patients with hip fractures demonstrated that 25% of patients suffered from undiagnosed DCM. Surgical decompression is the only form of treatment at present. It is shown to stop disease progression. However neurological recovery after surgery is often disappointing. There are no approved drug treatments for DCM. Alleviating the long-term disability caused by DCM represents an unmet clinical need. Recovery of leg and arm function, as well as an improvement in pain are the patient recovery priorities.

In DCM mechanical pressure on the spinal cord causes progressive loss of nerve cells and their processes as well as loss of myelin sheaths, the insulating layers of neurons formed by oligodendrocytes. Surgical decompression can halt disease progression, but there is limited natural spinal cord repair. Preclinical studies demonstrated that inhibition of PDE4 is able to stimulate a regenerative response, which is likely to benefit DCM: remyelination and axonal plasticity. Clinical studies using Ibudilast, a phosphodiesterase 4 inhibitor, have demonstrated beneficial effects in multiple sclerosis. The observed beneficial effects are likely to reflect regeneration-inducing and neuroprotective effects of Ibudilast in the human CNS.

The proposed trial is the first regenerative treatment for DCM, and potentially the first drug-based regenerative treatment for neurosurgical disease. It will mark an important milestone with regard to translation of preclinical findings into a clinical setting. The research questions have been designed to:

* Assess safety and tolerability of Ibudilast in patients undergoing surgery for DCM
* Assess efficacy of Ibudilast treatment in patients undergoing surgery for DCM
* Investigate disease mechanisms using

  * Advanced imaging techniques, including MRI
  * Gait analysis
* Explore the role of novel clinical outcome measures for studies investigating DCM

  * Clinical scales
* Inform the design of future drug trials for use in DCM
* Investigate the impact of DCM on carers

The following hypothesis will be addressed: Ibudilast improves recovery following surgical decompression of degenerative cervical myelopathy.

RECEDE-Myelopathy is a multi-centre, double blind, phase III randomised, placebo controlled trial assessing the use of Ibudilast as an adjuvant treatment to decompressive surgery for DCM involving up to 10 UK sites. A total of 362 participants will be recruited.

Each participant will be on trial for approximately 15 months (±21 days). There is a maximum 1 week interval from screening to randomisation and a maximum 1 week interval from randomisation to treatment commencement. Ibudilast treatment will start within 10 weeks prior to surgery and will continue for up to 24 weeks after surgery. Treatment will be halted 5 days prior to surgery and resumed at the previous maximum dose as soon as possible after two days since the operation. Participants will be taking Ibudilast for a maximum of 34 weeks; in case surgery is delayed beyond 10 weeks, post-surgery treatment will be shortened accordingly to keep the 34 weeks maximum treatment period. Participants will be followed up for a maximum of 12 months after surgery.

The trial aims to run in parallel to standard clinical care. The only difference between the trial pathway and the standard NHS pathway is the addition of a course of either Ibudilast or placebo, and the additional follow up.DCM is typically managed in the outpatient setting. Patients are referred to a surgeon for assessment and management. Patients often already have a diagnosis. Sometimes, an allied professional makes a diagnosis acutely and a same day, 'emergency' referral is made to the regional spinal centre. On occasion, such a situation predicates urgent surgery, but typically in such cases an outpatient appointment is made. Patients will therefore be identified from participating neurosurgical centres, typically via outpatient clinics but also the 'emergency' referrals. Screening of patients to determine eligibility for participation in the trial will be undertaken by the parent neurosurgical team according to the inclusion / exclusion criteria. Prior to screening, patients with DCM will be approached by a delegated member of the local trial team and given a patient information sheet (PIS) to take away and read in their own time. Patients will be advised to get in touch with the local trial team in order to address any questions that they may have on the contents of the PIS. If they decide to participate in the trial, they will be invited for a screening visit to provide a written informed consent and assess their eligibility for the trial as per inclusion/exclusion criteria described below.

Once informed consent is obtained, screening assessments will be performed in the same outpatient clinic visit.

Screening assessments to establish eligibility will include:

* Age
* Medical History including but not limited to

  * Neurological Disorder(s)
  * Respiratory Disorder(s)
  * Diabetes Mellitus
  * Psychiatric Disorder(s)
  * Smoking Status
* DCM characteristics

  * Symptoms
  * Length of DCM symptoms
  * Date of DCM diagnosis
  * MRI image findings and causative pathology
* Medication review, including allergy status
* Neurological examination
* mJOA assessment
* Laboratory Tests (FBC, LFT, E/U/C)
* Pregnancy test (serum beta HCG) - if female of childbearing potential (within 2 weeks of trial treatment start)
* ECG

Following screening assessments, trial-specific baseline assessments will be conducted, preferably on the same day.

* Demographics (weight (Kg), sex, ethnicity, date of birth)
* Employment status
* 30m walk test
* VAS pain
* SF-36
* EQ-5D/Health Resource usage
* Carer QoL (for sub-study)
* Review of potential AEs (starting from point of giving informed consent)
* A serum sample will be taken for PK studies Optional but highly desirable assessments
* GRASSP-Cervical Myelopathy
* SCIMv3
* NDI
* Quick-DASH

At the end of the visit, the dosing diary will be issued to the patient and instructed on how to use it. Participants' eligibility will be confirmed on receipt of results of the laboratory tests and they will be randomised to either Ibudilast or placebo. Participants will start treatment no later than 2 weeks after screening visit. One week after IMP delivery or collection, the local research team will make contact with the participant by telephone to ensure they have received the IMP and commenced their trial treatment. Any Adverse Events which may have occurred since consent will be documented in CRFs. Surgery will be performed, ideally, within 10 weeks after start of trial treatment.

Within 21 days prior to surgery, patients will have an outpatient clinic pre-operative visit and the following assessments will be performed:

* Laboratory Tests (FBC, LFT, E/U/C, TFTs)
* Assessment of any change to Medical or Drug history
* WHO performance status
* Neurological examination
* mJOA
* 30m walk test
* VAS pain
* SF-36
* EQ-5D/Health Resource usage
* Carer QoL (for sub-study)
* Review of AEs
* IMP compliance assessment (participant medication diary review and capsule count)
* Respiratory Physiology
* MRI
* Gait Lab (sub-study for Addenbrooke's only)
* A serum sample for PK studies will be taken Optional but highly desirable assessments
* GRASSP-Cervical Myelopathy
* SCIMv3
* NDI
* Quick-DASH

Intra-operative assessments

* Surgery details

  * Operation Title
  * Approach (Anterior, Posterior or Combined)
  * Instrumented Procedure?
  * Level(s) Treated
  * ASA
  * Intra-Operative Complications
* A CSF sample will be taken (if possible - optional)
* A paired serum sample for PK studies will be taken

Post-operative assessments on discharge (within 14 days after surgery)

* Neurological examination
* VAS Pain
* Adverse Events (including operative complications)
* IMP compliance assessment (participant medication diary review and capsule count)
* Further IMP will be dispensed

Optional but highly desirable assessments

• NDI

Follow Up assessments at 3 months post-surgery (±21 days)

* Laboratory Tests (FBC, LFT, E/U/C, TFTs)
* Neurological examination
* Medication review
* mJOA
* 30m walk test
* VAS pain
* SF-36
* Carer QoL (for sub-study)
* Review of AEs
* IMP compliance assessment (participant medication diary review and capsule count)
* A serum sample for PK studies will be taken Further IMP will be dispensed. Optional but highly desirable assessments
* GRASSP-Cervical Myelopathy
* NDI
* EQ-5D/Health Resource usage
* Quick-DASH
* Gait Lab (sub-study at Addenbrooke's only)

Follow Up assessments at 6 months post surgery (±21 days)

* Laboratory Tests (FBC, LFT, E/U/C, TFTs)
* Neurological examination
* Medication review
* mJOA
* 30m walk test
* VAS pain
* SF-36
* EQ-5D/Health Resource usage
* Carer QoL (for sub-study)
* Review of AEs
* IMP compliance (participant medication diary review and capsule count)
* Respiratory physiology
* MRI
* Gait lab (sub-study at Addenbrooke's only)
* A serum sample for PK studies will be taken Optional but highly desirable assessments
* GRASSP-Cervical Myelopathy
* SCIMv3
* NDI
* Quick-DASH

Follow Up assessments at 12 months post surgery (±21 days)

* Laboratory Tests (FBC, LFT, E/U/C, TFTs)
* Medication review
* Neurological examination
* mJOA
* 30m walk test
* VAS pain
* SF-36
* EQ-5D/Health Resource usage
* Carer QoL (for sub-study)
* Review of AEs
* A serum sample for PK studies will be taken Optional but highly desirable assessments
* GRASSP-Cervical Myelopathy
* NDI
* Quick-DASH

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from degenerative cervical myelopathy as per established criteria who have granted informed consent to participate in the trial
* Have a preoperative mJOA score ≥8 and ≤14
* Scheduled for first surgical decompression as part of usual NHS clinical practice

Exclusion Criteria:

* Previous surgery for DCM
* DCM symptoms due to cervical trauma (at the discretion of the investigator)
* Hypersensitivity to Ibudilast or any of the formulation components
* Evidence of acute hepatitis, clinically significant chronic hepatitis, or evidence of clinically significant impaired hepatic function through clinical and laboratory evaluation including ALP> 1.5x ULN; ALT or AST > 2x ULN; GGT > 3x ULN
* Active malignancy defined as history of invasive malignancy, except if the patient has received treatment and displayed no clinical signs and symptoms for at least five years
* Recent history (less than 3 years) of chemical substance dependency or significant psychosocial disturbance that may impact the outcome or study participation
* Female patients with child bearing potential who are unwilling or unable to use reliable methods of contraception
* Female patients who are pregnant, lactating or planning pregnancy during the course of the trial
* Inability to comply with study procedures, IMP regime or follow-up schedule
* Unable to take a gelatin based product
* Participation in another CTIMP or device within the past 30 days from the time of recruitment
* Functional disability from a commitment neurological disease that would mask the symptoms of DCM (at the discretion of the investigator). Including but not limited to stroke with residual disability, cerebellar ataxia, Parkinson's disease, symptomatic lumbar stenosis and multiple sclerosis
* Resting pulse < 50 bpm, SA or AV block, uncontrolled hypertension, or QTcF > 450 ms
* History of stomach or intestinal surgery or any other condition that could interfere with or is judged by the Investigator to interfere with absorption, distribution, metabolism, or excretion of study drug
* Unable to converse, read or write English at primary school level

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in modified Japanese Orthopaedic Association (mJOA) scale | From baseline to 6 months follow-up
  The mJOA is an 18-point clinician administered scale (0 worst to 18 best), which evaluates motor dysfunction in upper and lower extremities, loss of sensation and sphincter dysfunction.
Change in Visual Analogue Scale (VAS) neck pain | From baseline to 6 months follow-up
  VAS Neck pain is a 10cm horizontal line, on which a patient indicates their level of neck pain from 0 (no pain) to 10 (worst pain).

SECONDARY OUTCOMES:
PCS-SF36 | From baseline to 6 months follow-up
  SF-36 is a health and well-being questionnaire in which patient answers 36 multiple choice questions grouped under 11 sections. The answers to those questions are used to obtain the Physical Component Summary (PCS) of the SF-36 were lower scores indicate worse condition and higher score indicate better condition.
MCS-SF36 | From baseline to 6 months follow-up
  SF-36 is a health and well-being questionnaire in which patient answers 36 multiple choice questions grouped under 11 sections. The answers to those questions are used to obtain the Mental Component Summary (MCS) of the SF-36 were lower scores indicate worse condition and higher score indicate better condition.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Davies, MD, Principal Investigator — Cambridge University Hospital, Department of Neurosurgery
Locations (1):
- Addenbrooke's Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual participant's data will be shared with other researchers.

REFERENCES:
- [Background] Oh T, Lafage R, Lafage V, Protopsaltis T, Challier V, Shaffrey C, Kim HJ, Arnold P, Chapman J, Schwab F, Massicotte E, Yoon T, Bess S, Fehlings M, Smith J, Ames C. Comparing Quality of Life in Cervical Spondylotic Myelopathy with Other Chronic Debilitating Diseases Using the Short Form Survey 36-Health Survey. World Neurosurg. 2017 Oct;106:699-706. doi: 10.1016/j.wneu.2016.12.124. Epub 2017 Jan 5. PMID 28065875
- [Background] Davies BM, Mowforth OD, Smith EK, Kotter MR. Degenerative cervical myelopathy. BMJ. 2018 Feb 22;360:k186. doi: 10.1136/bmj.k186. No abstract available. PMID 29472200
- [Background] Nouri A, Tetreault L, Singh A, Karadimas SK, Fehlings MG. Degenerative Cervical Myelopathy: Epidemiology, Genetics, and Pathogenesis. Spine (Phila Pa 1976). 2015 Jun 15;40(12):E675-93. doi: 10.1097/BRS.0000000000000913. PMID 25839387
- [Background] Davies BM, Munro CF, Kotter MR. A Novel Insight Into the Challenges of Diagnosing Degenerative Cervical Myelopathy Using Web-Based Symptom Checkers. J Med Internet Res. 2019 Jan 11;21(1):e10868. doi: 10.2196/10868. PMID 30300137
- [Background] Chen LF, Tu TH, Chen YC, Wu JC, Chang PY, Liu L, Huang WC, Lo SS, Cheng H. Risk of spinal cord injury in patients with cervical spondylotic myelopathy and ossification of posterior longitudinal ligament: a national cohort study. Neurosurg Focus. 2016 Jun;40(6):E4. doi: 10.3171/2016.3.FOCUS1663. PMID 27246487
- [Background] Radcliff KE, Curry EP, Trimba R, Walker JB, Purtill JJ, Austin MS, Parvizi J, Vaccaro AR, Hilibrand AS, Albert TJ. High Incidence of Undiagnosed Cervical Myelopathy in Patients With Hip Fracture Compared With Controls. J Orthop Trauma. 2016 Apr;30(4):189-93. doi: 10.1097/BOT.0000000000000485. PMID 26562581
- [Background] Wu JC, Ko CC, Yen YS, Huang WC, Chen YC, Liu L, Tu TH, Lo SS, Cheng H. Epidemiology of cervical spondylotic myelopathy and its risk of causing spinal cord injury: a national cohort study. Neurosurg Focus. 2013 Jul;35(1):E10. doi: 10.3171/2013.4.FOCUS13122. PMID 23815246
- [Background] Wilson JR, Barry S, Fischer DJ, Skelly AC, Arnold PM, Riew KD, Shaffrey CI, Traynelis VC, Fehlings MG. Frequency, timing, and predictors of neurological dysfunction in the nonmyelopathic patient with cervical spinal cord compression, canal stenosis, and/or ossification of the posterior longitudinal ligament. Spine (Phila Pa 1976). 2013 Oct 15;38(22 Suppl 1):S37-54. doi: 10.1097/BRS.0b013e3182a7f2e7. PMID 23963005
- [Background] Kovalova I, Kerkovsky M, Kadanka Z, Kadanka Z Jr, Nemec M, Jurova B, Dusek L, Jarkovsky J, Bednarik J. Prevalence and Imaging Characteristics of Nonmyelopathic and Myelopathic Spondylotic Cervical Cord Compression. Spine (Phila Pa 1976). 2016 Dec 15;41(24):1908-1916. doi: 10.1097/BRS.0000000000001842. PMID 27509189
- [Background] Bednarik J, Kadanka Z, Dusek L, Kerkovsky M, Vohanka S, Novotny O, Urbanek I, Kratochvilova D. Presymptomatic spondylotic cervical myelopathy: an updated predictive model. Eur Spine J. 2008 Mar;17(3):421-431. doi: 10.1007/s00586-008-0585-1. Epub 2008 Jan 12. PMID 18193301
- [Background] Siivola SM, Levoska S, Tervonen O, Ilkko E, Vanharanta H, Keinanen-Kiukaanniemi S. MRI changes of cervical spine in asymptomatic and symptomatic young adults. Eur Spine J. 2002 Aug;11(4):358-63. doi: 10.1007/s00586-001-0370-x. Epub 2002 Feb 9. PMID 12193998
- [Background] Baptiste DC, Fehlings MG. Pathophysiology of cervical myelopathy. Spine J. 2006 Nov-Dec;6(6 Suppl):190S-197S. doi: 10.1016/j.spinee.2006.04.024. PMID 17097538
- [Background] Baron EM, Young WF. Cervical spondylotic myelopathy: a brief review of its pathophysiology, clinical course, and diagnosis. Neurosurgery. 2007 Jan;60(1 Supp1 1):S35-41. doi: 10.1227/01.NEU.0000215383.64386.82. PMID 17204884
- [Background] Kurokawa R, Murata H, Ogino M, Ueki K, Kim P. Altered blood flow distribution in the rat spinal cord under chronic compression. Spine (Phila Pa 1976). 2011 Jun;36(13):1006-9. doi: 10.1097/BRS.0b013e3181eaf33d. PMID 21192287
- [Background] Breig A, Turnbull I, Hassler O. Effects of mechanical stresses on the spinal cord in cervical spondylosis. A study on fresh cadaver material. J Neurosurg. 1966 Jul;25(1):45-56. doi: 10.3171/jns.1966.25.1.0045. No abstract available. PMID 5947047
- [Background] Karadimas SK, Laliberte AM, Tetreault L, Chung YS, Arnold P, Foltz WD, Fehlings MG. Riluzole blocks perioperative ischemia-reperfusion injury and enhances postdecompression outcomes in cervical spondylotic myelopathy. Sci Transl Med. 2015 Dec 2;7(316):316ra194. doi: 10.1126/scitranslmed.aac6524. PMID 26631633
- [Background] Yu WR, Liu T, Kiehl TR, Fehlings MG. Human neuropathological and animal model evidence supporting a role for Fas-mediated apoptosis and inflammation in cervical spondylotic myelopathy. Brain. 2011 May;134(Pt 5):1277-92. doi: 10.1093/brain/awr054. Epub 2011 Apr 13. PMID 21490053
- [Background] Fehlings MG, Ibrahim A, Tetreault L, Albanese V, Alvarado M, Arnold P, Barbagallo G, Bartels R, Bolger C, Defino H, Kale S, Massicotte E, Moraes O, Scerrati M, Tan G, Tanaka M, Toyone T, Yukawa Y, Zhou Q, Zileli M, Kopjar B. A global perspective on the outcomes of surgical decompression in patients with cervical spondylotic myelopathy: results from the prospective multicenter AOSpine international study on 479 patients. Spine (Phila Pa 1976). 2015 Sep 1;40(17):1322-8. doi: 10.1097/BRS.0000000000000988. PMID 26020847
- [Background] Fehlings MG, Wilson JR, Kopjar B, Yoon ST, Arnold PM, Massicotte EM, Vaccaro AR, Brodke DS, Shaffrey CI, Smith JS, Woodard EJ, Banco RJ, Chapman JR, Janssen ME, Bono CM, Sasso RC, Dekutoski MB, Gokaslan ZL. Efficacy and safety of surgical decompression in patients with cervical spondylotic myelopathy: results of the AOSpine North America prospective multi-center study. J Bone Joint Surg Am. 2013 Sep 18;95(18):1651-8. doi: 10.2106/JBJS.L.00589. PMID 24048552
- [Background] Tetreault LA, Skelly AC, Dettori JR, Wilson JR, Martin AR, Fehlings MG. Guidelines for the Management of Degenerative Cervical Myelopathy and Acute Spinal Cord Injury: Development Process and Methodology. Global Spine J. 2017 Sep;7(3 Suppl):8S-20S. doi: 10.1177/2192568217701715. Epub 2017 Sep 5. PMID 29164037
- [Background] Tetreault LA, Cote P, Kopjar B, Arnold P, Fehlings MG; AOSpine North America and International Clinical Trial Research Network. A clinical prediction model to assess surgical outcome in patients with cervical spondylotic myelopathy: internal and external validations using the prospective multicenter AOSpine North American and international datasets of 743 patients. Spine J. 2015 Mar 1;15(3):388-97. doi: 10.1016/j.spinee.2014.12.145. Epub 2014 Dec 27. PMID 25549860
- [Background] Alvin MD, Qureshi S, Klineberg E, Riew KD, Fischer DJ, Norvell DC, Mroz TE. Cervical degenerative disease: systematic review of economic analyses. Spine (Phila Pa 1976). 2014 Oct 15;39(22 Suppl 1):S53-64. doi: 10.1097/BRS.0000000000000547. PMID 25299260
- [Background] Witiw CD, Tetreault LA, Smieliauskas F, Kopjar B, Massicotte EM, Fehlings MG. Surgery for degenerative cervical myelopathy: a patient-centered quality of life and health economic evaluation. Spine J. 2017 Jan;17(1):15-25. doi: 10.1016/j.spinee.2016.10.015. Epub 2016 Oct 25. PMID 27793760
- [Background] Badran A, Davies BM, Bailey HM, Kalsi-Ryan S, Kotter MR. Is there a role for postoperative physiotherapy in degenerative cervical myelopathy? A systematic review. Clin Rehabil. 2018 Sep;32(9):1169-1174. doi: 10.1177/0269215518766229. Epub 2018 Apr 17. PMID 29663830
- [Background] Fehlings MG, Wilson JR, Karadimas SK, Arnold PM, Kopjar B. Clinical evaluation of a neuroprotective drug in patients with cervical spondylotic myelopathy undergoing surgical treatment: design and rationale for the CSM-Protect trial. Spine (Phila Pa 1976). 2013 Oct 15;38(22 Suppl 1):S68-75. doi: 10.1097/BRS.0b013e3182a7e9b0. PMID 23962993
- [Background] Dhillon RS, Parker J, Syed YA, Edgley S, Young A, Fawcett JW, Jeffery ND, Franklin RJ, Kotter MR. Axonal plasticity underpins the functional recovery following surgical decompression in a rat model of cervical spondylotic myelopathy. Acta Neuropathol Commun. 2016 Aug 23;4(1):89. doi: 10.1186/s40478-016-0359-7. PMID 27552807
- [Background] Karadimas SK, Erwin WM, Ely CG, Dettori JR, Fehlings MG. Pathophysiology and natural history of cervical spondylotic myelopathy. Spine (Phila Pa 1976). 2013 Oct 15;38(22 Suppl 1):S21-36. doi: 10.1097/BRS.0b013e3182a7f2c3. PMID 23963004
- [Background] Karadimas SK, Gatzounis G, Fehlings MG. Pathobiology of cervical spondylotic myelopathy. Eur Spine J. 2015 Apr;24 Suppl 2:132-8. doi: 10.1007/s00586-014-3264-4. Epub 2014 Mar 14. PMID 24626958
- [Background] Ito T, Oyanagi K, Takahashi H, Takahashi HE, Ikuta F. Cervical spondylotic myelopathy. Clinicopathologic study on the progression pattern and thin myelinated fibers of the lesions of seven patients examined during complete autopsy. Spine (Phila Pa 1976). 1996 Apr 1;21(7):827-33. doi: 10.1097/00007632-199604010-00010. PMID 8779013
- [Background] Nikulina E, Tidwell JL, Dai HN, Bregman BS, Filbin MT. The phosphodiesterase inhibitor rolipram delivered after a spinal cord lesion promotes axonal regeneration and functional recovery. Proc Natl Acad Sci U S A. 2004 Jun 8;101(23):8786-90. doi: 10.1073/pnas.0402595101. Epub 2004 Jun 1. PMID 15173585
- [Background] Syed YA, Baer A, Hofer MP, Gonzalez GA, Rundle J, Myrta S, Huang JK, Zhao C, Rossner MJ, Trotter MW, Lubec G, Franklin RJ, Kotter MR. Inhibition of phosphodiesterase-4 promotes oligodendrocyte precursor cell differentiation and enhances CNS remyelination. EMBO Mol Med. 2013 Dec;5(12):1918-34. doi: 10.1002/emmm.201303123. Epub 2013 Oct 21. PMID 24293318
- [Background] Gibson LC, Hastings SF, McPhee I, Clayton RA, Darroch CE, Mackenzie A, Mackenzie FL, Nagasawa M, Stevens PA, Mackenzie SJ. The inhibitory profile of Ibudilast against the human phosphodiesterase enzyme family. Eur J Pharmacol. 2006 May 24;538(1-3):39-42. doi: 10.1016/j.ejphar.2006.02.053. Epub 2006 Mar 13. PMID 16674936
- [Background] Smith FD, Langeberg LK, Cellurale C, Pawson T, Morrison DK, Davis RJ, Scott JD. AKAP-Lbc enhances cyclic AMP control of the ERK1/2 cascade. Nat Cell Biol. 2010 Dec;12(12):1242-9. doi: 10.1038/ncb2130. Epub 2010 Nov 21. PMID 21102438
- [Background] Cuadrado A, Nebreda AR. Mechanisms and functions of p38 MAPK signalling. Biochem J. 2010 Aug 1;429(3):403-17. doi: 10.1042/BJ20100323. PMID 20626350
- [Background] Pearse DD, Pereira FC, Marcillo AE, Bates ML, Berrocal YA, Filbin MT, Bunge MB. cAMP and Schwann cells promote axonal growth and functional recovery after spinal cord injury. Nat Med. 2004 Jun;10(6):610-6. doi: 10.1038/nm1056. Epub 2004 May 23. PMID 15156204
- [Background] Ji RR, Berta T, Nedergaard M. Glia and pain: is chronic pain a gliopathy? Pain. 2013 Dec;154 Suppl 1(0 1):S10-S28. doi: 10.1016/j.pain.2013.06.022. Epub 2013 Jun 20. PMID 23792284
- [Background] Kim HK, Kwon JY, Yoo C, Abdi S. The Analgesic Effect of Rolipram, a Phosphodiesterase 4 Inhibitor, on Chemotherapy-Induced Neuropathic Pain in Rats. Anesth Analg. 2015 Sep;121(3):822-828. doi: 10.1213/ANE.0000000000000853. PMID 26214551
- [Background] Guo CH, Bai L, Wu HH, Yang J, Cai GH, Wang X, Wu SX, Ma W. The analgesic effect of rolipram is associated with the inhibition of the activation of the spinal astrocytic JNK/CCL2 pathway in bone cancer pain. Int J Mol Med. 2016 Nov;38(5):1433-1442. doi: 10.3892/ijmm.2016.2763. Epub 2016 Sep 30. PMID 28025994
- [Background] Kostich W, Hamman BD, Li YW, Naidu S, Dandapani K, Feng J, Easton A, Bourin C, Baker K, Allen J, Savelieva K, Louis JV, Dokania M, Elavazhagan S, Vattikundala P, Sharma V, Das ML, Shankar G, Kumar A, Holenarsipur VK, Gulianello M, Molski T, Brown JM, Lewis M, Huang Y, Lu Y, Pieschl R, O'Malley K, Lippy J, Nouraldeen A, Lanthorn TH, Ye G, Wilson A, Balakrishnan A, Denton R, Grace JE, Lentz KA, Santone KS, Bi Y, Main A, Swaffield J, Carson K, Mandlekar S, Vikramadithyan RK, Nara SJ, Dzierba C, Bronson J, Macor JE, Zaczek R, Westphal R, Kiss L, Bristow L, Conway CM, Zambrowicz B, Albright CF. Inhibition of AAK1 Kinase as a Novel Therapeutic Approach to Treat Neuropathic Pain. J Pharmacol Exp Ther. 2016 Sep;358(3):371-86. doi: 10.1124/jpet.116.235333. Epub 2016 Jul 13. PMID 27411717
- [Background] Kim HK, Hwang SH, Oh E, Abdi S. Rolipram, a Selective Phosphodiesterase 4 Inhibitor, Ameliorates Mechanical Hyperalgesia in a Rat Model of Chemotherapy-Induced Neuropathic Pain through Inhibition of Inflammatory Cytokines in the Dorsal Root Ganglion. Front Pharmacol. 2017 Dec 4;8:885. doi: 10.3389/fphar.2017.00885. eCollection 2017. PMID 29255417
- [Background] Espirito-Santo RF, Meira CS, Costa RDS, Souza Filho OP, Evangelista AF, Trossini GHG, Ferreira GM, Velozo EDS, Villarreal CF, Pereira Soares MB. The anti-inflammatory and immunomodulatory potential of braylin: Pharmacological properties and mechanisms by in silico, in vitro and in vivo approaches. PLoS One. 2017 Jun 8;12(6):e0179174. doi: 10.1371/journal.pone.0179174. eCollection 2017. PMID 28594906
- [Background] Bao F, Fleming JC, Golshani R, Pearse DD, Kasabov L, Brown A, Weaver LC. A selective phosphodiesterase-4 inhibitor reduces leukocyte infiltration, oxidative processes, and tissue damage after spinal cord injury. J Neurotrauma. 2011 Jun;28(6):1035-49. doi: 10.1089/neu.2010.1575. Epub 2011 May 5. PMID 21355819
- [Background] Francischi JN, Yokoro CM, Poole S, Tafuri WL, Cunha FQ, Teixeira MM. Anti-inflammatory and analgesic effects of the phosphodiesterase 4 inhibitor rolipram in a rat model of arthritis. Eur J Pharmacol. 2000 Jul 7;399(2-3):243-9. doi: 10.1016/s0014-2999(00)00330-7. PMID 10884526
- [Background] Yamamoto S, Kurokawa R, Kim P. Cilostazol, a selective Type III phosphodiesterase inhibitor: prevention of cervical myelopathy in a rat chronic compression model. J Neurosurg Spine. 2014 Jan;20(1):93-101. doi: 10.3171/2013.9.SPINE121136. Epub 2013 Nov 8. PMID 24206033
- [Background] Rolan P, Hutchinson M, Johnson K. Ibudilast: a review of its pharmacology, efficacy and safety in respiratory and neurological disease. Expert Opin Pharmacother. 2009 Dec;10(17):2897-904. doi: 10.1517/14656560903426189. PMID 19929708
- [Background] Davies BM, McHugh M, Elgheriani A, Kolias AG, Tetreault LA, Hutchinson PJ, Fehlings MG, Kotter MR. Reported Outcome Measures in Degenerative Cervical Myelopathy: A Systematic Review. PLoS One. 2016 Aug 2;11(8):e0157263. doi: 10.1371/journal.pone.0157263. eCollection 2016. PMID 27482710
- [Background] Kalsi-Ryan S, Singh A, Massicotte EM, Arnold PM, Brodke DS, Norvell DC, Hermsmeyer JT, Fehlings MG. Ancillary outcome measures for assessment of individuals with cervical spondylotic myelopathy. Spine (Phila Pa 1976). 2013 Oct 15;38(22 Suppl 1):S111-22. doi: 10.1097/BRS.0b013e3182a7f499. PMID 23963009
- [Background] Kopjar B, Tetreault L, Kalsi-Ryan S, Fehlings M. Psychometric properties of the modified Japanese Orthopaedic Association scale in patients with cervical spondylotic myelopathy. Spine (Phila Pa 1976). 2015 Jan 1;40(1):E23-8. doi: 10.1097/BRS.0000000000000648. PMID 25341993
- [Background] Tetreault L, Nouri A, Kopjar B, Cote P, Fehlings MG. The Minimum Clinically Important Difference of the Modified Japanese Orthopaedic Association Scale in Patients with Degenerative Cervical Myelopathy. Spine (Phila Pa 1976). 2015 Nov;40(21):1653-9. doi: 10.1097/BRS.0000000000001127. PMID 26502097
- [Background] Fehlings MG, Martin AR, Tetreault LA, Aarabi B, Anderson P, Arnold PM, Brodke D, Burns AS, Chiba K, Dettori JR, Furlan JC, Hawryluk G, Holly LT, Howley S, Jeji T, Kalsi-Ryan S, Kotter M, Kurpad S, Kwon BK, Marino RJ, Massicotte E, Merli G, Middleton JW, Nakashima H, Nagoshi N, Palmieri K, Singh A, Skelly AC, Tsai EC, Vaccaro A, Wilson JR, Yee A, Harrop JS. A Clinical Practice Guideline for the Management of Patients With Acute Spinal Cord Injury: Recommendations on the Role of Baseline Magnetic Resonance Imaging in Clinical Decision Making and Outcome Prediction. Global Spine J. 2017 Sep;7(3 Suppl):221S-230S. doi: 10.1177/2192568217703089. Epub 2017 Sep 5. PMID 29164028
- [Background] Bogduk N, Govind J. Cervicogenic headache: an assessment of the evidence on clinical diagnosis, invasive tests, and treatment. Lancet Neurol. 2009 Oct;8(10):959-68. doi: 10.1016/S1474-4422(09)70209-1. PMID 19747657
- [Background] Schrot RJ, Mathew JS, Li Y, Beckett L, Bae HW, Kim KD. Headache relief after anterior cervical discectomy: post hoc analysis of a randomized investigational device exemption trial: clinical article. J Neurosurg Spine. 2014 Aug;21(2):217-22. doi: 10.3171/2014.4.SPINE13669. Epub 2014 May 16. PMID 24836655
- [Background] Segerdahl M. Pain outcome variables--a never ending story? Pain. 2011 May;152(5):961-962. doi: 10.1016/j.pain.2011.03.008. No abstract available. PMID 21439731
- [Background] MacDowall A, Skeppholm M, Robinson Y, Olerud C. Validation of the visual analog scale in the cervical spine. J Neurosurg Spine. 2018 Mar;28(3):227-235. doi: 10.3171/2017.5.SPINE1732. Epub 2017 Dec 15. PMID 29243996
- [Background] Parker SL, Godil SS, Shau DN, Mendenhall SK, McGirt MJ. Assessment of the minimum clinically important difference in pain, disability, and quality of life after anterior cervical discectomy and fusion: clinical article. J Neurosurg Spine. 2013 Feb;18(2):154-60. doi: 10.3171/2012.10.SPINE12312. Epub 2012 Nov 23. PMID 23176164
- [Background] Auffinger BM, Lall RR, Dahdaleh NS, Wong AP, Lam SK, Koski T, Fessler RG, Smith ZA. Measuring surgical outcomes in cervical spondylotic myelopathy patients undergoing anterior cervical discectomy and fusion: assessment of minimum clinically important difference. PLoS One. 2013 Jun 24;8(6):e67408. doi: 10.1371/journal.pone.0067408. Print 2013. PMID 23826290
- [Background] Tetreault LA, Kopjar B, Vaccaro A, Yoon ST, Arnold PM, Massicotte EM, Fehlings MG. A clinical prediction model to determine outcomes in patients with cervical spondylotic myelopathy undergoing surgical treatment: data from the prospective, multi-center AOSpine North America study. J Bone Joint Surg Am. 2013 Sep 18;95(18):1659-66. doi: 10.2106/JBJS.L.01323. PMID 24048553
- [Background] Martin AR, Aleksanderek I, Cohen-Adad J, Tarmohamed Z, Tetreault L, Smith N, Cadotte DW, Crawley A, Ginsberg H, Mikulis DJ, Fehlings MG. Translating state-of-the-art spinal cord MRI techniques to clinical use: A systematic review of clinical studies utilizing DTI, MT, MWF, MRS, and fMRI. Neuroimage Clin. 2015 Dec 4;10:192-238. doi: 10.1016/j.nicl.2015.11.019. eCollection 2016. PMID 26862478
- [Background] Floeth FW, Galldiks N, Eicker S, Stoffels G, Herdmann J, Steiger HJ, Antoch G, Rhee S, Langen KJ. Hypermetabolism in 18F-FDG PET predicts favorable outcome following decompressive surgery in patients with degenerative cervical myelopathy. J Nucl Med. 2013 Sep;54(9):1577-83. doi: 10.2967/jnumed.112.113183. Epub 2013 Aug 5. PMID 23918736
- [Background] Bhagavatula ID, Bhat DI, Sasidharan GM, Mishra RK, Maste PS, Vilanilam GC, Sathyaprabha TN. Subclinical respiratory dysfunction in chronic cervical cord compression: a pulmonary function test correlation. Neurosurg Focus. 2016 Jun;40(6):E3. doi: 10.3171/2016.3.FOCUS1647. PMID 27246486
- [Background] Ellis RJ, Ng YS, Zhu S, Tan DM, Anderson B, Schlaug G, Wang Y. A Validated Smartphone-Based Assessment of Gait and Gait Variability in Parkinson's Disease. PLoS One. 2015 Oct 30;10(10):e0141694. doi: 10.1371/journal.pone.0141694. eCollection 2015. PMID 26517720
- [Background] Raknim P, Lan KC. Gait Monitoring for Early Neurological Disorder Detection Using Sensors in a Smartphone: Validation and a Case Study of Parkinsonism. Telemed J E Health. 2016 Jan;22(1):75-81. doi: 10.1089/tmj.2015.0005. Epub 2015 Aug 24. PMID 26302109
- [Background] Mourcou Q, Fleury A, Franco C, Klopcic F, Vuillerme N. Performance Evaluation of Smartphone Inertial Sensors Measurement for Range of Motion. Sensors (Basel). 2015 Sep 15;15(9):23168-87. doi: 10.3390/s150923168. PMID 26389900
- [Background] Sanftner LM, Gibbons JA, Gross MI, Suzuki BM, Gaeta FC, Johnson KW. Cross-species comparisons of the pharmacokinetics of ibudilast. Xenobiotica. 2009 Dec;39(12):964-77. doi: 10.3109/00498250903254340. PMID 19925385
- [Background] DeYoung DZ, Heinzerling KG, Swanson AN, Tsuang J, Furst BA, Yi Y, Wu YN, Moody DE, Andrenyak DM, Shoptaw SJ. Safety of Intravenous Methamphetamine Administration During Ibudilast Treatment. J Clin Psychopharmacol. 2016 Aug;36(4):347-54. doi: 10.1097/JCP.0000000000000511. PMID 27269956
- [Background] Goodman AD, Gyang T, Smith AD 3rd. Ibudilast for the treatment of multiple sclerosis. Expert Opin Investig Drugs. 2016 Oct;25(10):1231-7. doi: 10.1080/13543784.2016.1221924. Epub 2016 Aug 22. PMID 27501293
- [Background] Barkhof F, Hulst HE, Drulovic J, Uitdehaag BM, Matsuda K, Landin R; MN166-001 Investigators. Ibudilast in relapsing-remitting multiple sclerosis: a neuroprotectant? Neurology. 2010 Mar 30;74(13):1033-40. doi: 10.1212/WNL.0b013e3181d7d651. Epub 2010 Mar 3. PMID 20200338
- [Background] van Waesberghe JH, Kamphorst W, De Groot CJ, van Walderveen MA, Castelijns JA, Ravid R, Lycklama a Nijeholt GJ, van der Valk P, Polman CH, Thompson AJ, Barkhof F. Axonal loss in multiple sclerosis lesions: magnetic resonance imaging insights into substrates of disability. Ann Neurol. 1999 Nov;46(5):747-54. doi: 10.1002/1531-8249(199911)46:53.3.co;2-w. PMID 10553992
- [Background] Pirko I, Johnson A, Gamez J, Macura SI, Rodriguez M. Disappearing "T1 black holes" in an animal model of multiple sclerosis. Front Biosci. 2004 May 1;9:1222-7. doi: 10.2741/1322. PMID 14977539
- [Background] Kwok YH, Swift JE, Gazerani P, Rolan P. A double-blind, randomized, placebo-controlled pilot trial to determine the efficacy and safety of ibudilast, a potential glial attenuator, in chronic migraine. J Pain Res. 2016 Oct 31;9:899-907. doi: 10.2147/JPR.S116968. eCollection 2016. PMID 27826212
- [Background] Johnson JL, Kwok YH, Sumracki NM, Swift JE, Hutchinson MR, Johnson K, Williams DB, Tuke J, Rolan PE. Glial Attenuation With Ibudilast in the Treatment of Medication Overuse Headache: A Double-Blind, Randomized, Placebo-Controlled Pilot Trial of Efficacy and Safety. Headache. 2015 Oct;55(9):1192-208. doi: 10.1111/head.12655. Epub 2015 Sep 14. PMID 26367865
- [Background] Rolan P, Gibbons JA, He L, Chang E, Jones D, Gross MI, Davidson JB, Sanftner LM, Johnson KW. Ibudilast in healthy volunteers: safety, tolerability and pharmacokinetics with single and multiple doses. Br J Clin Pharmacol. 2008 Dec;66(6):792-801. doi: 10.1111/j.1365-2125.2008.03270.x. PMID 19032723
- [Background] Yoon H, Cho HY, Lee YB. Determination of ibudilast in human serum by high-performance liquid chromatography for pharmacokinetic study. Biomed Chromatogr. 2010 Mar;24(3):324-8. doi: 10.1002/bmc.1293. PMID 19629961
- [Background] Nagata K, Ohashi T, Abe J, Morita M, Inoue A. Cervical myelopathy in elderly patients: clinical results and MRI findings before and after decompression surgery. Spinal Cord. 1996 Apr;34(4):220-6. doi: 10.1038/sc.1996.41. PMID 8963966
- [Background] Helmy A, Guilfoyle MR, Carpenter KL, Pickard JD, Menon DK, Hutchinson PJ. Recombinant human interleukin-1 receptor antagonist in severe traumatic brain injury: a phase II randomized control trial. J Cereb Blood Flow Metab. 2014 May;34(5):845-51. doi: 10.1038/jcbfm.2014.23. Epub 2014 Feb 26. PMID 24569690
- [Background] Tetreault L, Wilson JR, Kotter MR, Nouri A, Cote P, Kopjar B, Arnold PM, Fehlings MG. Predicting the minimum clinically important difference in patients undergoing surgery for the treatment of degenerative cervical myelopathy. Neurosurg Focus. 2016 Jun;40(6):E14. doi: 10.3171/2016.3.FOCUS1665. PMID 27246484
- [Background] Sculpher M, Drummond M, Buxton M. The iterative use of economic evaluation as part of the process of health technology assessment. J Health Serv Res Policy. 1997 Jan;2(1):26-30. doi: 10.1177/135581969700200107. PMID 10180650
- [Background] Ramsey SD, Willke RJ, Glick H, Reed SD, Augustovski F, Jonsson B, Briggs A, Sullivan SD. Cost-effectiveness analysis alongside clinical trials II-An ISPOR Good Research Practices Task Force report. Value Health. 2015 Mar;18(2):161-72. doi: 10.1016/j.jval.2015.02.001. PMID 25773551
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] van Hout B, Janssen MF, Feng YS, Kohlmann T, Busschbach J, Golicki D, Lloyd A, Scalone L, Kind P, Pickard AS. Interim scoring for the EQ-5D-5L: mapping the EQ-5D-5L to EQ-5D-3L value sets. Value Health. 2012 Jul-Aug;15(5):708-15. doi: 10.1016/j.jval.2012.02.008. Epub 2012 May 24. PMID 22867780